CLINICAL TRIAL: NCT06333080
Title: The Effect of Adherence to Oral Semaglutide on Glycaemic Control in People With Type 2 Diabetes Treated With Metformin (DIACRON) - An Open-label Clinical Trial
Brief Title: The Effect of Adherence to Oral Semaglutide on Glycaemic Control in People With Type 2 Diabetes Treated With Metformin
Acronym: DIACRON
Status: Recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Peter Vestergaard, Professor and Endocrinologist, Aalborg University Hospital
Other Study IDs: N-20220017
Record Dates: First submitted 2024-02-05; First posted 2024-03-27 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Treatment Adherence and Compliance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: People with dysregulated type 2 diabetes on metformin treatment, which are naïve to second line antidiabetic treatment. These participants will be started on oral semaglutide, as a second line antidiabetic treatment, in addition to their treatment with metformin. The participants will be started on 3mg and the dose increased according to the label. The oral semaglutide will be administered once daily.

SUMMARY:
The objective of the trial is to investigate the effect of adherence to oral semaglutide dosing instructions on glycaemic control in people with type 2 diabetes, which are dysregulated on metformin and naïve to second line antidiabetic treatment.

DETAILED DESCRIPTION:
The trial is a prospective non-interventional clinical trial with a duration of 12 weeks and will be conducted at Steno Diabetes Center North Denmark (SDCN)/the Endocrinology Outpatient Clinic, Aalborg University Hospital.

The participants of this non-interventional clinical trial are people with T2D, which are dysregulated on metformin and naïve to second line antidiabetic treatment. As these patients do not have glycaemic control despite treat-ment with metformin and lifestyle interventions, the next recommended step in the treatment, according to current guidelines, is to add a second line antidiabetic to the treatment. As the treatment, according to guidelines, should be individualised, only patients which would start treatment with oral semaglutide independently of this trial are eligible for trial inclusion.

The trial period starts with the first visit to the trial site and ends 12 weeks later with the second visit to the trial site. A CGM baseline of each participant is collected prior to oral semaglutide initiation, corresponding to the two first weeks of the trial period. After oral semaglutide initiation, CGM data, physical activity, time of dosing, and water volume intake at dosing time are collected throughout the remaining trial period. The participants are asked to report occurrences of nausea and vomiting including time, duration, and severity (using a scale from 0-10, as previously described). In addition, the participants are asked to register time of breakfast at 3 time periods of the clinical trial.

The patient-reported adherence and satisfaction of the diabetes treatment is assessed using the TRIM-D, which is a questionnaire consisting of 28 questions, divided into five subcategories: treatment burden, daily life, diabetes management, compliance, and psychological health. The participants are asked to electronically answer the TRIM-D questionnaire at the start and end of the trial. The TRIM-D questionnaire is used in the validated Danish version. Data on health belief is obtained by asking the participants to answer the questionnaire developed by Given, et al. and adapted by Becker and Janz. The participants will furthermore be asked to answer a questionnaire on social support, developed by Sarason, et al. The questionnaires on health belief and social support are translated to Danish.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes for at least 1 year.
* HbA1c of 53-75 mmol/mol at ???.
* Treated with metformin for at least 1 year.
* Can understand and read Danish.
* Can use a smartphone, as well as the devices used in the clinical trial.
* Signed informed consent.

Exclusion Criteria:

* HbA1c value recorded less than 3 months prior to inclusion in trial.
* Current or prior treatment with other glucose-lowering medications than metformin.
* Cardiovascular disease or kidney disease which would indicate use of other second line treatments such as SGLT2 inhibitors or s.c. GLP1 receptor agonists (see also current guidelines https://endocrinology.dk/nbv/diabetes-melitus/behandling-og-kontrol-af-type-2-diabetes/).
* Other types of diabetes than type 2 diabetes.
* Participation in other trials.
* Pregnancy or breastfeeding.
* Known retinopathy.
* Known allergy to semaglutide.
* Major surgery planned during the trial period.
* Cancer diagnosis within five years prior to inclusion.
* Personal or family history of medullary thyroid carcinoma.
* Multiple endocrine neoplasia syndrome type 2.
* Conditions, which the investigators deem to render the participant unfit for inclusion in the trial, including a physical or cognitive inability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included participants must have type 2 diabetes, which is dysregulated on metformin and be naïve to second line antidiabetic treatment. Participants are regarded as dysregulated if a HbA1c of 53-75 mmol/mol has been recorded 3 months prior to trial inclusion and again at the first visit. As the participants do not have glycaemic control, the next step in the treatment is to initiate a second line antidiabetic treatment, which in this clinical trial is oral semaglutide. Thus, eligible participants for this study should have a second line antidiabetic treatment added to their metformin treatment, regardless of participation in this study. The participants will continue their metformin treatment and treatment with oral semaglutide will be initiated two weeks after trial start.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Time-in-Range (TIR) | Change from baseline to three-month assessment
  Change from baseline to end-of-study in time-in-range (TIR) derived from CGM calculated in accordance with the International Consensus on Use of Continuous Glucose Monitoring.

SECONDARY OUTCOMES:
Pre-dose Fasting | Time (minutes) elapsed from last registered food intake to registered medication intake.
  Pre-dose fasting, defined as the time elapsed from last food intake in the evening to dosing time.
Post-dose Fasting | Time (minutes) elapsed from registered medication intake to registered time of breakfast (start).
  Post-dose fasting, defined as time elapsed from dosing time to time of breakfast.
Occurrence of nausea or vomiting | Reported during the entire trial duration, three months.
  Occurrence of nausea or vomiting incl. timing, duration, and severity. Nausea and vomiting severity are reported on a scale from 0-10 with 0 being no nausea/vomiting and 10 being the worst imaginable nausea/vomiting, similar to the scale of nausea severity described by Leere, et al.
Water Intake at Dosing Time | Collected during the entire trial duration, three months.
  Volume of water intake at dosing time.
Treatment-Related Impact Measure for Diabetes (TRIM-D) | Change from baseline to end of trial (three-month assessment).
  Patient-reported satisfaction and adherence of treatment reported as the total score of the treatment-related impact measure for diabetes (TRIM-D).

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center North Denmark, Aalborg, Denmark

REFERENCES:
- [Derived] Holdt-Caspersen NS, Dethlefsen C, Hejlesen O, Christiansen E, Hangaard S, Vestergaard P, Jensen MH. Effect of Adherence to Oral Semaglutide on Glycemic Control in People With Type 2 Diabetes Treated With Metformin: Protocol for an Open-Label Clinical Trial. JMIR Res Protoc. 2025 Sep 23;14:e64899. doi: 10.2196/64899. PMID 40986866